CLINICAL TRIAL: NCT03981341
Title: Impact of Estrogen + Estradiol Receptor Alpha Modulator Therapy on Oxidative Stress in Post-menopausal Women With and Without Sleep Apnea
Acronym: Alpha MenoX
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Collaborators: V Joseph (Unknown); C Minville (Unknown); C Rheaume (Unknown)
Responsible Party: Principal Investigator, Frédéric Sériès, Director IUCPQ sleep clinic, Laval University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IUCPQ220519
Record Dates: First submitted 2019-05-22; First posted 2019-06-10 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Sleep Apnea; Post Menopausal; Oxidative Stress
Keywords: sleep apnea; post menopausal; oxidative stress
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — bazedoxifene

STUDY DESIGN:
Intervention Model Description: Open label treatment for 3 months in two parallel groups (post menopausal women without and with sleep apnea)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Post menopausal sleep apnea (Experimental): Post menopausal women with severe sleep apnea
  Interventions: Drug: Duavive (0.45 estrogens mg and 20 mg bazedoxifene)
- Post menopausal non sleep apnea (Experimental): Post menopausal women without sleep apnea
  Interventions: Drug: Duavive (0.45 estrogens mg and 20 mg bazedoxifene)

INTERVENTIONS:
Drug: Duavive (0.45 estrogens mg and 20 mg bazedoxifene) — Drug given for 3 months in each participant

SUMMARY:
One of the most likely mechanisms explaining the sleep apnea (SA)-induced increase in metabolic syndrome is the oxidative stress (OS) induced by intermittent hypoxia (IH). There are clear-cut signs of OS in postmenopausal women that may be further enhanced by SA. In rats exposed to IH, an estradiol receptor alpha agonist decreases the level of OS markers. The aims of this study are to compare OS in apneic and non-apneic postmenopausal women and to demonstrate that OS will improve after 3 months of treatment with ER alpha agonists (Duavive) in apneic post-menopausal women.

DETAILED DESCRIPTION:
Sleep apnoea (SA) is highly prevalent in general population. It is a sex-specific respiratory disease with a lower incidence in women than in men but it increases after menopause. SA and nocturnal intermittent hypoxia (IH) predict the risks of metabolic syndrome independently of obesity, and in patients without comorbidities, SA is associated with insulin resistance. One of the most likely mechanisms explaining the SA-induced increase in metabolic syndrome is the oxidative stress (OS) induced by IH. There are clear-cut signs of OS in postmenopausal women that may be further enhanced by SA resulting in an increased activity of the sympathetic system as well as damages in adipose tissue, blood vessels, and in the liver. Estradiol is a potent antioxidant hormone. Recent experiments conducted in Dr Joseph laboratory demonstrated that in ovariectomized female rats exposed to IH, an ER alpha agonist decreases the level of "Advanced Oxidation Protein Products", prevents excessive mitochondrial ROS production, and the increase of arterial blood pressure. Oestrogens combined with a tissue-specific estradiol receptor modulators (bazedoxifene) are approved and available in Canada (Duavive) for the treatment of vasomotor symptoms and prevention of osteoporosis associated with menopause. The aims of this study are to compare OS in apneic and non-apneic postmenopausal women and to demonstrate that OS will improve after 3 months of treatment with ER alpha agonists (Duavive) in apneic post-menopausal women. 18 newly diagnosed women with untreated severe SA and 18 without SA will be recruited from the sleep clinic. Eligible subjects will be post-menopausal non-smoking women aged 30 to 65 years with a BMI less/equal to 35 kg.m-2, apnoea + hypopnea index < 15/h (non SA group) or ≥ 30/h (SA group) on a polysomnographic recording. The study will be a prospective comparative trial. Following completion of baseline measurements, subjects will receive 1 tablet of Duavive (0.45 estrogens mg and 20 mg bazedoxifene) daily for 3 months. A follow-up phone call will be completed monthly, and side effects will be recorded. All measurements will be repeated after 3 months of Duavive. The main outcome is the levels of Advanced Oxidation Protein Products and malondialdehyde as a reflect of cellular oxidative damages. The investigators will also measure plasmatic activity of superoxide dismutase and serum nitrite + nitrate levels. Secondary outcomes are related to metabolic (anthropometric variables, biologic markers of glucose homeostasis, lipid profiles, orexin-A and liver function), cardiac health (arterial blood pressure, 24-h heart rate variability to measure cardiac autonomic function) and quality of life. Analysis: Differences between results obtained in each condition will be analysed using ANOVA. Statistical significance will be considered at p<0.05. Considering the changes in OS observed with hormonal therapy in post-menopausal women and those observed with SA treatment, the sample size was determined to be able to demonstrate a 30 % difference in OS between SA and non-apneic women following 3 month of treatment with Duavive with alpha =0.05, 80% power analysis and a 20% drop-out rate. New avenues in postmenauposal hormonal therapy may have a huge impact on morbidity/mortality and a drug therapy should be more easily accepted that CPAP to reach this goal. These results should open the door to an RCT aimed at quantifying benefits of such treatment on metabolic syndrome features.

ELIGIBILITY:
Inclusion Criteria:

* post-menopausal women
* aged 45 to 65 years
* BMI less/equal 35 kg.m-2,
* apnoea + hypopnea index (AHI) < 15/h (non SA group) or ≥ 30/h (SA group) on a polysomnographic recording,
* 90% of AHI associated with obstructive events,
* regular exercise, dietary and sleep habits
* free of sleep debt (insomnia, reported habitual sleep time > 6 h/night),
* stable medical condition.

Exclusion Criteria:

* clinically significant diurnal somnolence requiring immediate treatment in SA patients,
* nocturnal hypoventilation (% sleep time below 90% SaO2 > 10 %, PaCO2 > 45 mmHg),
* use of hormonal therapy,
* use of any medication with a respiratory depressant effect (narcotics),
* contraindication to the dug used in the protocol

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — post menopausal women
Enrollment: 36 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
oxidative stress | Changes between baseline and after 3 months drug treatment
  Advanced Oxidation Protein Products

SECONDARY OUTCOMES:
glucose homeostasis | Changes between baseline and after 3 months drug treatment
  HOMA-IR
total cholesterol | Changes between baseline and after 3 months drug treatment
  serum cholesterol
triglycerides | Changes between baseline and after 3 months drug treatment
  serum triglycerides
aspartate aminotransferase (AST) | Changes between baseline and after 3 months drug treatment
  serum aspartate aminotransferase
gamma-glutamyl transferase (∂-GT) | Changes between baseline and after 3 months drug treatment
  serum gamma-glutamyl transferase
Orexin-A | Changes between baseline and after 3 months drug treatment
  Orexin-A
C-reactive protein | Changes between baseline and after 3 months drug treatment
  serum C-reactive protein
arterial blood pressure | Changes between baseline and after 3 months drug treatment
  resting arterial blood pressure
heart rate variability | Changes between baseline and after 3 months drug treatment
  24-holter

CONTACTS AND LOCATIONS:
Locations (1):
- IUCPQ, Québec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laouafa S, Ribon-Demars A, Marcouiller F, Roussel D, Bairam A, Pialoux V, Joseph V. Estradiol Protects Against Cardiorespiratory Dysfunctions and Oxidative Stress in Intermittent Hypoxia. Sleep. 2017 Aug 1;40(8). doi: 10.1093/sleep/zsx104. PMID 28633495
- [Background] Barrera J, Chambliss KL, Ahmed M, Tanigaki K, Thompson B, McDonald JG, Mineo C, Shaul PW. Bazedoxifene and conjugated estrogen prevent diet-induced obesity, hepatic steatosis, and type 2 diabetes in mice without impacting the reproductive tract. Am J Physiol Endocrinol Metab. 2014 Aug 1;307(3):E345-54. doi: 10.1152/ajpendo.00653.2013. Epub 2014 Jun 17. PMID 24939737
- [Background] Xue B, Zhao Y, Johnson AK, Hay M. Central estrogen inhibition of angiotensin II-induced hypertension in male mice and the role of reactive oxygen species. Am J Physiol Heart Circ Physiol. 2008 Sep;295(3):H1025-H1032. doi: 10.1152/ajpheart.00021.2008. Epub 2008 Jul 3. PMID 18599599
- [Background] de Lima AM, Franco CM, de Castro CM, Bezerra Ade A, Ataide L Jr, Halpern A. Effects of nasal continuous positive airway pressure treatment on oxidative stress and adiponectin levels in obese patients with obstructive sleep apnea. Respiration. 2010;79(5):370-6. doi: 10.1159/000227800. Epub 2009 Jul 3. PMID 19590157